CLINICAL TRIAL: NCT03479736
Title: A Self-Controlled Case Series Study of Fluoroquinolones Exposure and Collagen-related Serious Adverse Events
Brief Title: A Study of Fluoroquinolones Exposure and Collagen-Related Serious Adverse Events
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108453; RRA-19796 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Retinal Detachment; Achilles Tendon; Aneurysm, Dissecting
MeSH Terms: conditions — Retinal Detachment; Aortic Dissection | interventions — Fluoroquinolones

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Cohort 1: Participants with Achilles Tendon Rupture (ATR): Participants will be defined as having ATR if they receive a diagnosis for ATR as well as one of the following procedures: tenotomy or primary ruptured Achilles Tendon (AT) repair (with or without graft) within 7 days of diagnosis. Index will be based on the earlier date of diagnosis or procedure. Participants with ATR, and exposures to Fluoroquinolone (FQ) or any of the other antibiotics or febrile illness not treated with antibiotic, within a defined study period and at least 1 year of continuous enrollment prior to the event will be included. It will use data from 3 databases, which are Truven CCAE and Medicare (Supplemental) and Optum ClinFormatics (Optum).
  Interventions: Drug: Oral Fluoroquinolones (FQ); Drug: Other Antibiotics; Other: Febrile Illness Not Treated with Antibiotics Will be Analyzed as an Exposure
- Cohort 2: Participants with Retinal Detachment (RD): Participants will be defined as having a RD if they received a diagnosis of RD and a procedure for RD, e.g.: sclera buckle, vitrectomy, retinopexy, retinal cryotherapy, silicone oil fill, air gas fluid exchange or pneumatic retinopexy, within 14 days of index. Index will be defined as the earlier date of diagnosis or procedure. Participants with RD, and exposures to FQ or any of the other antibiotics or febrile illness not treated with antibiotic, within a defined study period and at least 1 year of continuous enrollment prior to the event will be included. It will use data from 3 databases, which are Truven CCAE and Medicare (Supplemental) and Optum ClinFormatics (Optum).
  Interventions: Drug: Oral Fluoroquinolones (FQ); Drug: Other Antibiotics; Other: Febrile Illness Not Treated with Antibiotics Will be Analyzed as an Exposure
- Cohort 3: Participants with Aortic Aneurysm & Dissection (AAD): Participants will be defined as having AAD if they received a primary diagnosis for aortic aneurysm, aortic rupture or dissection and have also received an aortic repair surgical procedure concurrently to the AAD diagnosis, in an inpatient or emergency department (ED) setting. Index will be defined as the earlier date of diagnosis or procedure. Participants with AAD, and exposures to FQ or any of the other antibiotics or febrile illness not treated with antibiotic, within a defined study period and at least 1 year of continuous enrollment prior to the event will be included. It will use data from 3 databases, which are Truven CCAE and Medicare (Supplemental) and Optum ClinFormatics (Optum).
  Interventions: Drug: Oral Fluoroquinolones (FQ); Drug: Other Antibiotics; Other: Febrile Illness Not Treated with Antibiotics Will be Analyzed as an Exposure

INTERVENTIONS:
Drug: Oral Fluoroquinolones (FQ) — Participants will not receive any intervention as a part of this study. The FQ include all oral forms of FQ (24-hours extended release tablets, extended release tablets, oral solution, oral suspension, oral tablet, pack). The drugs included are ciprofloxacin, gatifloxacin, gemifloxacin, levofloxacin, moxifloxacin, norfloxacin, ofloxacin.
Drug: Other Antibiotics — Participants will not receive any intervention as a part of this study. Other antibiotics include amoxicillin, azithromycin, trimethoprim and trimethroprim/sulfamethoxazole.
Other: Febrile Illness Not Treated with Antibiotics Will be Analyzed as an Exposure — Febrile illness not treated with antibiotics is defined as: concurrent diagnoses of viral disease with concurrent fever, and no concurrent prescription for any antibiotic during the 60-day period before and after the first date of viral disease diagnosis; or a diagnosis of influenza with no concurrent inpatient admission during the 60-day period pre- or post-influenza diagnosis, and no prescription for any antibiotics during the 60-day period pre- or post-influenza diagnosis.

SUMMARY:
The purpose of this study is to evaluate whether there is an increased risk of achilles tendon rupture (ATR), retinal detachment (RD) or aortic aneurysm and dissection (AAD) following exposure to fluoroquinolone (FQ) or other antibiotics (amoxicillin, azithromycin, trimethoprim and trimethroprim/sulfamethoxazole) or febrile illness not treated with antibiotics, using a study design that minimizes the impact of confounders not usually captured in health services databases such as heredity or smoking.

ELIGIBILITY:
Inclusion Criteria:

* Have evidence of at least 1 instance of Achilles Tendon Rupture (ATR) or Retinal Detachment (RD) or Aortic Aneurysm and Dissection (AAD)
* Have at least 1 exposure to Fluoroquinolones or any of the other antibiotics (amoxicillin, azithromycin, trimethoprim and trimethroprim/sulfamethoxazole) or febrile illness not treated with antibiotic
* Have at least 1 year of continuous enrollment with pharmacy benefits prior to the ATR, RD or AAD

Exclusion Criteria:

ATR, AAD and RD cohorts:

- Participants who experience the index event while within a time-at-risk window for more than one exposure type. (The exposure types in this study include FQ as a class, amoxicillin, azithromycin, trimethoprim, trimethroprim/sulfamethoxazole, and febrile illness not treated with antibiotics. Events while within a time-at-risk window of two or more exposure types cannot be associated with any one exposure. Participants are therefore excluded from the study)

For ATR and AAD cohorts:

* Have inherited disorders of connective tissue, specifically: Ehlers-Danlos syndrome, epidermolysis bullosa, Marfan syndrome, osteogenesis imperfecta
* Have an ATR or AAD event prior to index, during the 1-year pre-index period

For RD cohort:

* Have cataract surgery prior to index
* Have iridotomy or iridectomy prior to index

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants with Achilles Tendon Rupture (ATR) or Retinal Detachment (RD) or Aortic Aneurysm and Dissection (AAD), and exposures to Fluoroquinolones (FQ) or any of the other antibiotics or febrile illness not treated with antibiotic, within a defined study period and at least 1 year of continuous enrollment prior to the event.
Sampling Method: Non-Probability Sample
Enrollment: 117911 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Number of Events Resulting From Collagen-Related Disorders Achilles Tendon Rupture (ATR), Retinal Detachment (RD) and Aortic Aneurysm and Dissection (AAD) by Exposure to Fluoroquinolones (FQ) | Approximately up to 6 years
  Participants will be having ATR if they receive a diagnosis for ATR and 1 of the following: tenotomy/primary ruptured AT repair (with/without graft) within 7 days of diagnosis. Participants will be having RD if they receive a diagnosis of RD and a procedure for RD, e.g.: sclera buckle, vitrectomy, retinopexy, retinal cryotherapy, silicone oil fill, air gas fluid exchange or pneumatic retinopexy, within 14 days of index (earlier date of diagnosis/procedure). Participants will be having AAD if they receive a diagnosis for aortic aneurysm, aortic rupture/dissection and an aortic repair surgical procedure concurrently to it, in an inpatient/ED setting. The FQ include all oral forms of FQ (ciprofloxacin, gatifloxacin, gemifloxacin, levofloxacin, moxifloxacin, norfloxacin, ofloxacin). Relative risk of RD, ATR, and AAD between periods of exposure and non-exposure to FQ will be assessed using number of events. Temporal associations between RD, ATR or AAD and exposure to FQ will be estimated.
Number of Events Resulting From Collagen-Related Disorders ATR, RD and AAD by Exposure to Other Antibiotics | Approximately up to 6 years
  Other antibiotics includes amoxicillin, azithromycin, trimethoprim and trimethroprim/sulfamethoxazole. Relative risk of RD, ATR, and AAD between periods of exposure and non-exposure to other antibiotics will be assessed using number of events. Temporal associations between RD, ATR or AAD and exposure to other antibiotics will be estimated.
Number of Events Resulting From Collagen-Related Disorders ATR, RD and AAD by Febrile Illness Not Treated With Antibiotics | Approximately up to 6 years
  Febrile illness not treated with antibiotics is defined as: concurrent diagnoses of viral disease with concurrent fever, and no concurrent prescription for any antibiotic during the 60-day period before and after the first date of viral disease diagnosis; or a diagnosis of influenza with no concurrent inpatient admission during the 60-day period pre- or post-influenza diagnosis, and no prescription for any antibiotics during the 60-day period pre- or post-influenza diagnosis. Relative risk of RD, ATR, and AAD between periods of exposure and non-exposure to febrile illness not treated with antibiotics will be assessed using number of events. Temporal associations between RD, ATR or AAD and febrile illness not treated with antibiotics (analyzed as an exposure) will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Janssen Investigative Site, Titusville, New Jersey, United States

REFERENCES:
- [Derived] Londhe AA, Holy CE, Weaver J, Fonseca S, Villasis-Keever A, Fife D. Risk of retinal detachment and exposure to fluoroquinolones, common antibiotics, and febrile illness using a self-controlled case series study design: Retrospective analyses of three large healthcare databases in the US. PLoS One. 2022 Oct 6;17(10):e0275796. doi: 10.1371/journal.pone.0275796. eCollection 2022. PMID 36201545
- [Derived] Londhe AA, Holy CE, Weaver J, Fonseca S, Villasis A, Fife D. Risk of aortic aneurysm and dissection following exposure to fluoroquinolones, common antibiotics, and febrile illness using a self-controlled case series study design: Retrospective analyses of three large healthcare databases in the US. PLoS One. 2021 Aug 16;16(8):e0255887. doi: 10.1371/journal.pone.0255887. eCollection 2021. PMID 34398907